CLINICAL TRIAL: NCT00288496
Title: Mechanical Bowel Preparation for Elective Colorectal Surgery. A Multicenter Randomized Study
Brief Title: Mechanical Bowel Preparation for Elective Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ikazia Hospital, Rotterdam (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POCON trial
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2006-02-08 (Estimated); Status verified 2000-04

CONDITIONS: Anastomotic Dehiscence in Colorectal Surgery
Keywords: mechanical bowel preparation, colorectal surgery, anastomotic dehiscence

INTERVENTIONS:
Drug: polyethylene glycol bowel lavage solution

SUMMARY:
Mechanical bowel preparation (MBP) is common practice in elective colorectal surgery. In recent literature the value of MBP is subject of discussion. We conducted a multicenter, randomized study with the goal of comparing outcome of elective colorectal resections and primary anastomoses with and without mechanical bowel preparation in terms of anastomotic leakage and other septic complications.

Within the setting of a multicenter randomized trial,1433 patients were randomized before elective colorectal surgery to receive either MBP or to have no MBP but a normal meal on the day before operation. The primary endpoint was anastomotic leakage. Secondary endpoints were septic complications (wound infection, urinary infection, pneumonia, pelvic abscesses), fascia dehiscence and death.

The incidence of anastomotic leakage was similar in both groups: 5.1% in patients without MBP versus 4.9% in patients with MBP (p=0.93; 95% confidence interval for the difference (no MBP minus MBP) ranges from -2.3% tot +2.7%). There were no significant differences in other septic complications, fascia dehiscence, or mortality. Fecal contamination, number of days until resumption of a normal diet, and duration of hospital stay were similar in both groups.

This study shows that elective colorectal surgery can be safely done without MBP. Therefore, MBP should be abandoned in elective colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criterion was elective colorectal surgery with primary anastomosis

Exclusion Criteria:

Exclusion criteria were an acute laparotomy, laparoscopic colorectal surgery, contraindications for the use of mechanical bowel preparation, an a priori deviating (ileo) stoma, and age less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400
Dates: Start 1998-04; Study Completion 2004-02

PRIMARY OUTCOMES:
The primary endpoint of the study was anastomotic failure.

SECONDARY OUTCOMES:
Secondary endpoints were septic complications (wound infection, urinary infection, pneumonia, pelvic abscesses), fascia dehiscence and death.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ME Contant, PhD, Principal Investigator — Ikazia Hospital
Locations (1):
- Caroline Contant, Rotterdam, Montessoriweg 1, Netherlands

REFERENCES:
- [Derived] Contant CM, Hop WC, van't Sant HP, Oostvogel HJ, Smeets HJ, Stassen LP, Neijenhuis PA, Idenburg FJ, Dijkhuis CM, Heres P, van Tets WF, Gerritsen JJ, Weidema WF. Mechanical bowel preparation for elective colorectal surgery: a multicentre randomised trial. Lancet. 2007 Dec 22;370(9605):2112-7. doi: 10.1016/S0140-6736(07)61905-9. PMID 18156032